CLINICAL TRIAL: NCT05894863
Title: Smart Flex Stent System for the Treatment Long Femoropopliteal Artery Lesions: the SAFARI Study
Brief Title: Smart Flex Stent System for the Treatment Long Femoropopliteal Artery Lesions
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: RenJi Hospital (Other)
Collaborators: Xuanwu Hospital, Beijing (Other); Second Affiliated Hospital of Soochow University (Other); First Affiliated Hospital of Zhejiang University (Other); First People's Hospital of Hangzhou (Other); Qingdao Haici Hospital (Other); Liyuan Hospital of Tongji Medical College, Huazhong University of Science and Technology (Other); Fudan University (Other); Dongfang Hospital Beijing University of Chinese Medicine (Other); Xiamen Cardiovascular Hospital, Xiamen University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: The SAFARI Study
Record Dates: First submitted 2023-05-31; First posted 2023-06-08 (Actual); Last update posted 2023-06-08 (Actual); Status verified 2023-05

CONDITIONS: Peripheral Arterial Disease
Keywords: Femoropopliteal lesions; Patency
MeSH Terms: conditions — Peripheral Arterial Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Smart flex stent group (Experimental): Smart flex stent will be used for patients with femoropopliteal lesions receiving endovascular treatment.
  Interventions: Device: Smart flex stent

INTERVENTIONS:
Device: Smart flex stent — Smart flex stent will be used for femoropopliteal occlusive lesions.

SUMMARY:
This study aims to evaluate the effectiveness and safety of the Smart flex stent system in treating long femoropopliteal native lesions.

DETAILED DESCRIPTION:
One hundred twenty patients with lesion lengths longer than 15 cm will be included. Patients will be invited for a follow-up visit at 1, 6, 12, and 24-month post-procedure. The primary effectiveness endpoint of the study is the primary patency at 12 months. The primary safety endpoint is freedom of major adverse events (MAEs) at 12 months. Secondary endpoints include acute procedure success rate; primary patency rate at 1, 6, and 24 months; freedom from TLR at 1-, 6-, 12, and 24-month follow-up; primary and secondary sustained clinical improvements at 1-, 6-, 12- and 24-month follow-up; Freedom of MAEs at 1-, 6-,12- and 24- month follow-up; change of quality of life at 1-, 6-,12- and 24- month follow-up.

ELIGIBILITY:
Inclusion Criteria:

1. The patient presented a score from 2 to 5 following Rutherford classification
2. The patient is willing to comply with specified follow-up evaluations at the specified times
3. The patient is >18 years old
4. Patient understands the nature of the procedure and provides written informed consent before enrolment in the study
5. The patient has a projected life expectancy of at least 24 months
6. Before enrolment, the guidewire has crossed the target lesion
7. Target lesion length ≧150mm by angiographic estimation
8. Stenosis > 50% or occlusion in the femoropopliteal artery
9. There is angiographic evidence of patent distal popliteal artery and at least one distal runoff to the foot

Exclusion Criteria:

1. Previous bypass surgery or stenting in the target vessel
2. Patients who exhibit acute intraluminal thrombus at the target lesion vessel
3. Patients with known hypersensitivity or contraindication to any of the following medications: Nitinol-titanium, antiplatelet therapy, anticoagulants, or thrombolytics therapy
4. Pregnant women or Female patients with potential childbearing
5. Use of thrombectomy, atherectomy, or laser devices during the procedure
6. Untreated inflow disease of the ipsilateral pelvic arteries (more than 50% stenosis or occlusion
7. The patient is currently participating in another investigational drug or device study that has not reached the primary endpoint.
8. Significant renal dysfunction (Serum creatinine >2.0mg/dl)
9. Patient with Known allergy to contrast media

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2023-05-31 (Actual); Primary Completion 2026-01-02 (Estimated); Study Completion 2027-01-02 (Estimated)

PRIMARY OUTCOMES:
Primary patency | 12-month
  Primary patency is freedom from clinically directed target lesion revascularization (CD-TLR) and from Duplex ultrasound-derived binary restenosis (defined as peak systolic velocity ratio ≧2.5).
Freedom of major adverse events (MAEs) | 12-month
  Major adverse events(MAEs) is defined as index limb amputation above the ankle, clinically directed target lesion revascularization(CD-TLR), or all-cause death.

SECONDARY OUTCOMES:
Acute procedure success | 72-hour within procedure
  Acute procedure success is defined as technique success ( the achievement of final residual diameter stenosis <30% for stent and <50% for angioplasty or atherectomy by angiography at the end of the procedure and without flow-limiting arterial dissection or hemodynamically significant trans-lesional pressure gradient <10 mm Hg for endovascular revascularization ) and freedom form major adverse events.
Primary patency | 24-month
  Primary patency is freedom from clinically directed target lesion revascularization (CD-TLR) and from Duplex ultrasound-derived binary restenosis (defined as peak systolic velocity ratio ≧2.5).
Freedom from clinically directed target lesion revascularization | 24-month
  Patients without clinically directed target lesion revascularization
Freedom of major adverse events (MAEs) | 24-month
  Major adverse events(MAEs) is defined as index limb amputation above the ankle, clinically directed target lesion revascularization(CD-TLR), or all-cause death.
Primary sustained clinical improvement | 24-month
  Primary sustained clinical improvement is defined as an upward shift on the Rutherford classification to a level of claudication without the need for repeated TLR in surviving patients without the need for unplanned amputation.
Vasc quality of life score | 24-month
  Change of Vasc quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Meng Ye, M.D., Principal Investigator — Department of Vascular Surgery, Renji Hospital, School of Medicine, Shanghai Jiaotong University
Locations (1):
- Renji Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No